CLINICAL TRIAL: NCT04157959
Title: A Phase I, Single-Center, Open-Label Study to Evaluate Pharmacodynamics of Drug-Drug Interaction Between SHR4640 and Febuxostat in Patients With Hyperuricemia
Brief Title: The Drug-Drug Interaction of SHR4640 and Febuxostat in Patients With Hyperuricemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHR4640-104
Record Dates: First submitted 2019-11-04; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR4640 (Experimental): SHR4640 dose1 Oral Tablet Day1~Day14 qd,Febuxostat dose2 Oral Tablet Day8 and Day14 qd.
  Interventions: Drug: SHR4640 dose1; Drug: Febuxostat dose2
- Febuxostat (Experimental): Febuxostat dose2 Oral Tablet Day1 and Day14 qd, SHR4640 dose1 Oral Tablet Day8~Day14 qd.
  Interventions: Drug: SHR4640 dose1; Drug: Febuxostat dose2

INTERVENTIONS:
Drug: SHR4640 dose1 — Tablet,dose1,QD
Drug: Febuxostat dose2 — Tablet,dose2,QD

SUMMARY:
The objective of the study is to assess the pharmacodynamic properties of drug-drug of SHR4640 and Febuxostat interaction in patients with Hyperuricemia.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a body mass index ≥18 and ≤30 kg/m2;
2. Screening sUA value ≥8mg/dl;
3. Subject has no clinically relevant abnormalities in vital signs, ECG, physical examination，imaging examination or safety laboratory values.

Exclusion Criteria:

1. Subject known or suspected of being sensitive to the study drugs or its ingredient；
2. ALT、AST、TBIL>ULN;
3. History of kidney stones or screening kidney stones by B-ultrasound；
4. History of malignancy；
5. History of xanthinuria；
6. Donated blood（≥400ml）within 3 months prior to screening or received transfusion of blood。

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of SHR4640 and Febuxostat from plasma | Day1 to Day 14
Area under the plasma concentration versus time curve (AUC) of SHR4640 and Febuxostat from plasma | Day1 to Day 14

SECONDARY OUTCOMES:
Apparent terminal half-life (t1/2) of SHR4640 and Febuxostat from plasma | Day1 to Day 14
Number of Participants With Adverse Events (AEs) and Serious Adverse Events | Clinical significant changes from Day-21 up to Day 29
  Laboratory indicators, 12-lead electrocardiogram (ECG), physical examination,vital signs, adverse events (NCI-CTC AE 5.0), etc.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of QingDao University, Qingdao, Shandong, China

REFERENCES:
- [Derived] Wang C, Yu Q, Jiang X, Deng Y, Sun F, Li X, Tao Y, Lin P, Ma Y, Zhu Y, Li C, Cao Y. A Drug-Drug Interaction Study of a Novel Selective Urate Reabsorption Inhibitor, SHR4640, and Xanthine Oxidase Inhibitor, Febuxostat, in Patients With Primary Hyperuricemia. J Clin Pharmacol. 2023 Feb;63(2):239-249. doi: 10.1002/jcph.2159. Epub 2022 Oct 20. PMID 36131360